CLINICAL TRIAL: NCT00891254
Title: Randomized Study of Long-term Follow-up of Incisional Hernia Repaired With Intraperitoneal Mesh Versus On-lay Mesh Repair
Brief Title: Long-term Follow-up of Incisional Hernia Repaired With Intraperitoneal Mesh
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Principal Investigator, MARCELO A. BELTRAN, M.D., DIGESTIVE SURGEON, Cirujanos la Serena
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLS-2904009-03
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; Intraperitoneal mesh repair; On-lay repair; Prosthetic mesh; First repair (no recurrent hernia will be included); Recurrence; Complications
MeSH Terms: conditions — Incisional Hernia; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Intraperitoneal repair (Active Comparator): Patients with incisional hernia, 5 cm in diameter or with an area of 25 cm2, submitted to elective surgery
  Interventions: Device: Implant of a prosthetic mesh
- 2. On-Lay repair (Active Comparator): Patients with incisional hernia, with a diameter of 5 cm or an area of 25 cm2, submitted to elective surgery
  Interventions: Device: Implant of a prosthetic mesh

INTERVENTIONS:
Device: Implant of a prosthetic mesh — A prosthetic mesh will be implanted either intraperitoneally or in the on-lay (supra-fascial) position depending on the arm of the study

SUMMARY:
The intraperitoneal repair has been proven safe for the repair of incisional hernia and is accepted, together with the subfascial or retromuscular repair as the "gold-standard" for the repair of incisional hernia. However no studies have convincingly proven that this approach is better than the on-lay repair.

The authors believe that the intraperitoneal repair performs better than the on-lay repair for incisional hernia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incisional hernia 5 cm of diameter or with an area of 25 square cm (cm2)
* First repair
* Older than 35 years of age and younger than 75 years of age
* Both genders
* Any BMI
* Only upper abdominal midline incisional hernias (supraumbilical)
* Patients submitted only to elective repair

Exclusion Criteria:

* Recurrent incisional hernia
* Emergency surgery
* Hernias with a diameter higher than 5 cm or more than 25 cm2 of area
* Lower midline abdominal incisional hernias
* Other hernias rather than midline incisional hernias
* Non-incisional hernias

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Long-term recurrence | 5 years

SECONDARY OUTCOMES:
Short-term complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO A BELTRAN, M.D., Principal Investigator — Hospital de La Serena
Locations (1):
- Hospital de La Serena, La Serena, Coquimbo Region, Chile